CLINICAL TRIAL: NCT04438408
Title: National Survey on Care Pathway and Quality of Life in Patients With Severe Asthma According to Their Phenotype.
Acronym: 2ndsouffle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0285
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Asthma Chronic; Severe Asthma
Keywords: Severe Asthma; Th2 phenotype; Care pathway; Quality of life
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe asthma patient: Adult patients (≥ 18 years) with diagnosis of severe asthma for at least 12 months
  Interventions: Other: questionaires

INTERVENTIONS:
Other: questionaires — patients will answer to questionnaires on the quality of life and the control of the asthmatic disease as well as the therapeutic observance.

SUMMARY:
The SECOND SOUFFLE survey focuses on aspects of care and quality of life in a period when the landscape of severe asthma is changing in the context of biotherapies. Moreover survey on care pathway and quality of life of the asthmatic severe population according to their phenotype have never been done. It is likely to bring results in a relatively fast time, results that can lead to guide the criteria collected in RAMSES a national severe asthma cohort and future research tracks of this cohort.

DETAILED DESCRIPTION:
The Th2 phenotype corresponds to severe asthmatic patients eligible for new subcutaneous targeted asthma therapies, which can bring about a real improvement in symptoms and quality of life. No data are available on the proportion of this patient population since the advent of biotherapies, as well as the impact on quality of life and pathway by phenotype.

The survey will be conducted using a collection of data on a dedicated questionnaire including validated questionnaires on the quality of life and the control of the asthmatic disease as well as the therapeutic observance.

The objectives of the survey are to estimate the phenotypic profile distribution of severe asthmatic patients and the proportion currently treated by biotherapies as well as the impact of the pathology on the clinical profile and quality of life of patients with severe asthma.

Investigative pulmonologists selected from university or general hospitals or from private practice will propose to their eligible patients to participate in the study. Patients informed and not opposed to participating will complete, at the end of the consultation, the dedicated questionnaire pre-filled by the pulmonologist (for the medical data required for phenotypic stratification). The questionnaires will be collected from the centers and the data centralized to establish the database. Analyzes will be done in order to stratify the populations according to their phenotype and to analyze the data globally and by subgroup.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe asthma for at least 12 months confirmed by a respiratory physicians and meeting the ATS / ERS definition,
* Social insured patient,
* Patient given the non-opposition

Exclusion Criteria:

* Patient participating in a therapeutic clinical trial
* Patient opposing participation in this study
* Patient with reading and comprehension difficulties not allowing him to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed diagnosis of severe asthma for at least 12 months
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Stratification of severe asthmatics in 3 phenotypes | 12 months
  The severe asthmatics patients will stratified in 3 phenotypes groups: Th2 phenotype with biotherapy, Th2 phenotype without biotherapy and non-Th2 phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Didier Alain, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No